CLINICAL TRIAL: NCT06552234
Title: Open-label Phase II Efficacy Study of Repotrectinib in Frail (PS ≥2) and/or Elderly Patients With ROS1-rearranged Advanced NSCLC
Brief Title: Phase II Efficacy Study of Repotrectinib in Frail and/or Elderly Patients With ROS1-rearranged Advanced NSCLC
Acronym: REPOROS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Groupe Francais De Pneumo-Cancerologie (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REPOROS GFPC 04-2023; 2023-509073-23-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-01; First posted 2024-08-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: NSCLC Stage IV; NSCLC, Stage III
Keywords: tyrosine-kinase inhibitors; Frail patients; Elderly patients; ROS1 rearrangements; resistance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — repotrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Repotrectinib treatment (Experimental): patient treated by Repotrectinib until progression or unacceptable toxicity
  Interventions: Drug: Repotrectinib

INTERVENTIONS:
Drug: Repotrectinib — Repotrectinib 160 mg BID, until progression or unacceptable toxicity

SUMMARY:
ROS1 rearrangements are rare, accounting for only 1-2% of NSCLC cases, but have been associated with response to ROS1 inhibitors, such as crizotinib and entrectinib. However, many patients develop resistance to the tyrosine-kinase inhibitors (TKIs), creating a need for new treatments.

Repotrectinib is a new-generation TKI designed against ROS1 or NTRK rearranged malignancies (Drilon 2018). Early phase clinical data support activity of repotrectinib in patients with NSCLC harboring such gene rearrangements (TRIDENT-1 study), but there are limited evidence in frail populations, such as poor performance status patients and/or elderly patients, who are classically excluded from clinical trials or underrepresented.

The present study aims to assess the activity and tolerability of repotrectinib in frail (PS ≥2) and/or elderly patients with ROS1-rearranged advanced NSCLC.

DETAILED DESCRIPTION:
This is a national, multicenter, phase II, prospective, open label, non-randomized, interventional study.

Frail (PS≥2) and/or elderly patients (≥70 years) with histologically/cytologically proven stage IV or stage III non-eligible to local treatment NSCLC harboring an ROS1 gene rearrangement treated by Repotrectinib (160 mg twice a day (BID), until progression or unacceptable toxicity) in first or any line.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are defined as patients with

  * Eastern Cooperative Oncology Group (ECOG) PS ≥ 2 at the time of inclusion and/or
  * Age ≥ 70 years
* Age ≥ 18 years
* Histologically or cytologically confirmed diagnosis of locally advanced or metastatic NSCLC harboring an ROS1 gene rearrangement as by any nucleic acid-based diagnostic testing method (e.g., next-generation sequencing [NGS], Sanger sequencing, reverse transcription-polymerase chain reaction), Break-apart fluorescence in situ hybridization (FISH) or Immunohistochemistry (IHC) (confirmed by NGS or qPCR test).
* Willing and able to provide written institutional review board (IRB)/institutional ethics committee-approved Informed Consent.
* At least 1 measurable target lesion according to RECIST (v1.1). CNS-only measurable disease as defined by RECIST (v1.1) is allowed.
* Prior cytotoxic chemotherapy for advanced or metastatic disease is allowed. At the time of starting treatment with repotrectinib, at least 14 days or 5 half-lives (whichever is shorter) must have elapsed after discontinuation of prior cytotoxic chemotherapy (or at least 42 days for prior nitrosoureas, mitomycin C, and liposomal doxorubicin) and all side effects from prior treatments must have resolved to grade ≤ _1 (CTCAE Version 5.0 with the exception of alopecia.
* Prior immunotherapy (e.g., anti-PD-1, anti-PDL1, anti-TIM3, anti-OX40) is allowed. At the time of starting treatment with repotrectinib, at least 14 days must have elapsed after discontinuation of prior immunotherapy treatment and all immune-related side effects from prior treatments must have resolved to grade ≤ _1.
* No prior ROS1 TKI is allowed for the TKI naïve cohort.
* Prior ROS1 TKI is allowed for the TKI pretreated cohort (max 30% of patients). At least 7 days or 5 half-lives (whichever is shorter) must have elapsed since completion of treatment with the last ROS1i prior to starting treatment with repotrectinib for subjects enrolling into the TKI-pretreated expansion cohorts. All side effects from prior treatments with ROS1i must have resolved to grade ≤ _1 prior to starting treatment with repotrectinib.

  * Prior ROS1i allowed include crizotinib, ceritinib, lorlatinib, brigatinib, entrectinib, ensartinib, cabozantinib.
* Subjects with symptomatic CNS metastases and/or asymptomatic leptomeningeal carcinomatosis are eligible.
* Life expectancy ≥3 months
* Subject affiliated to an appropriate social security system
* Adequate hematologic and end-organ function, defined by the following laboratory

  * ANC ≥ 1500 /mm3 without granulocyte colony-stimulating factor support
  * Lymphocyte count ≥ 500/mm3
  * Platelet count ≥ 100,000/mm3 without transfusion
  * Hemoglobin ≥ 9.0 g/dL. Patients may be transfused to meet this criterion.
  * INR or aPTT ≤ 1.5, upper limit of normal (ULN)
  * This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be receiving a stable dose.
  * ASAT, ALAT, and alkaline phosphatase ≤ 2.5xULN, with the following exceptions:
  * Patients with documented liver metastases: ASAT and/or ALAT ≤ 5xULN
  * Patients with documented liver or bone metastases: alkaline phosphatase < 5xULN
  * Serum bilirubin ≤1.25xULN
  * Patients with known Gilbert disease who have serum bilirubin level ≤ 3xULN may be enrolled.
  * Calculated creatinine clearance (CRCL) ≥ 45 mL/min
* Adequate method of contraception during the treatment period

  * For Females:

All women of childbearing potential (WOCBP) must agree to avoid pregnancy during the study and must use a highly effective method of contraception during study treatment with repotrectinib and for at least 2 months following the final dose.

Highly effective contraceptive methods consist of prior sterilization, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), injectable or implantable contraceptives and abstinence.

Hormonal contraception must begin 7 days prior to the first dose of study treatment.

Due to a potential loss of effectiveness of hormonal contraceptives caused by interaction with study intervention, if WOCBP use hormonal contraceptives (including oral hormonal contraceptives), they must use either another form of non-hormonal highly effective contraception or a reliable barrier method.

Female subjects must refrain from egg donation from screening through at least 2 months after the last dose of study drug.

* For Males:

Male participants with WOCBP partners must use latex condoms during treatment with repotrectinib and for 4 months following the final dose even if the participant has undergone a successful vasectomy or if the partner is pregnant or breastfeeding.

Male subjects must refrain from sperm donation from screening through at least 4 months after the last dose of study drug

Exclusion Criteria:

* Malignancies other than NSCLC within 2 years prior to inclusion, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS ≥ 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous-cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)
* Patients with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible only if they are negative for HBV DNA. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA.
* Active tuberculosis
* Severe infections within 2 weeks prior to inclusion, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction, or cerebrovascular accident within 3 months prior to inclusion, unstable arrhythmias, or unstable angina
* Major surgical procedure other than for diagnosis within 28 days prior to inclusion or anticipation of need for a major surgical procedure during the course of the study
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications.
* Patients with illnesses or conditions that interfere with their capacity to understand follow and/or comply with study procedures.
* Concurrent participation in any therapeutic clinical trial
* Patient deprived of liberty or placed under the authority of a tutor or a curator
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2031-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) according to RECIST v1.1. | From the date of first treatment administration until the date of disease progression or death if patient died before progression) or the introduction of a new treatment, which ever occurs earlier, assessed up to 7 years
  ORR defined as the proportion of patients who achieved a complete or partial response according to RECIST v1.1 from the date of first treatment administration until disease progression or death if patient died before progression or the introduction of a new treatment assessed by blinded independent central review.
  Tumor assessments will be performed at Screening, every 2 Months during the first year then every 3 months thereafter until documented progression, death or the introduction of a new treatment.
  Patients who discontinue treatment for reasons other than radiographic disease progression per RECIST v1.1 (toxicity, symptomatic deterioration) will continue scheduled tumor assessments until radiographic disease progression per RECIST v1.1, withdrawal of consent, death, or study termination by the co-Sponsors, whichever occurs first

SECONDARY OUTCOMES:
Progression free survival (PFS) by masked, independent central review | From the date of first treatment administration until the date of disease progression (or death if patient died before progression), which ever occurs earlier, assessed up to 7 years
  Independent central review of progression free survival (PFS) from Repotrectinib initiation, defined as the time from first dose of Repotrectinib to first documentation of objective disease progression (RECIST v1.1) or to death from any cause. Patients lost to follow-up will be censored as the last date of radiological assessment without progression.
  Tumor assessments will be performed at Screening, every 2 Months during the first year then every 3 months thereafter until documented progression, death or the introduction of a new treatment.
  Patients who discontinue treatment for reasons other than radiographic disease progression per RECIST v1.1 (e.g., toxicity, symptomatic deterioration) will continue scheduled tumor assessments until radiographic disease progression per RECIST v1.1, withdrawal of consent, death, or study termination by the co-Sponsors, whichever occurs first.
Disease control rate (DCR) by masked, independent central review | From the date of first treatment administration until the date of disease progression (or death if patient died before progression), which ever occurs earlier, assessed up to 7 years
  DCR, defined as the proportion of patients who achieved a complete response (CR) or partial response (PR) or stable disease (SD) according to RECIST v1.1 assessed by BICR.
  Tumor assessments will be performed at Screening, every 2 Months during the first year then every 3 months thereafter until documented progression, death or the introduction of a new treatment.
  Patients who discontinue treatment for reasons other than radiographic disease progression per RECIST v1.1 (e.g., toxicity, symptomatic deterioration) will continue scheduled tumor assessments until radiographic disease progression per RECIST v1.1, withdrawal of consent, death, or study termination by the co-Sponsors, whichever occurs first.
Intracranial ORR (ic-ORR) by masked, independent central review | From the date of first treatment administration until the date of disease progression (or death if patient died before progression), which ever occurs earlier, assessed up to 7 years
  ic-ORR, defined as the proportion of patients who achieved CR or PR in measurable brain metastases based on RECIST 1.1 criteria
Overall survival (OS) | From the date of first treatment administration until the date of death from any cause, assessed up to 7 years
  OS, defined as the time from first dose of Repotrectinib until death from any cause. Patients lost to follow-up will be censored at the last date known to be alive.
  OS will be evaluated every 3 months (until death or lost to follow-up) in patients who:
  * Discontinue the study treatment due to disease progression
  * Discontinue the study treatment due to an unacceptable toxicity or any other reason, and who start a new therapy
  * Reach the End-of-study Time Point.
Toxicities occurring during either the induction or maintenance treatment in terms of kind, grade, time of onset, reversibility, according to NCI-CTCAE v5.0 criteria | From the date of first treatment administration up to 30 days after the last dose of study treatment
  Proportion (%) of patients with any adverse event (AE) and number of events for all AEs, all serious AEs (SAEs) and all AEs of grade ≥3 according to the National Cancer Institute (NCI) Common terminology criteria for adverse events (CTCAE) v5.0 criteria.
Duration of response (DOR) assessed in patients who had an objective response as determined by the investigator using RECIST v1.1 | From the date of first documented objective response (CR or PR) until disease progression or death, which ever occurs earlier, assessed up to 7 years
  DOR, defined as the time from the first documented objective response (CR or PR) until disease progression or death, whichever occurs first.
Time to deterioration in lung-related symptoms | From the date of inclusion to the date the patient's score on the EORTC QLQ C30 or QLQ-LC13 shows a ≥10-point increase above baseline, assessed up to 7 years
  Time to deterioration in lung-related symptoms, defined as the time from inclusion to the time the patient's score on the EORTC QLQ C30 or QLQ-LC13 shows a ≥10-point increase above baseline in each of the following EORTC-transformed scores for cough, dyspnea (single item), dyspnea (multi-item subscale) and chest pain. Patients lost to follow-up without previous QOL deterioration will be censored at the last EORTC assessment date.
  QoL/PRO questionnaires may be filled out up until D1 every 8 weeks ±7 days during the first year, then every 12 weeks ±7 days thereafter at Progression.
Time to deterioration in quality of life | From the date of inclusion to the date the patient's score on the EQ-5D-3L utility score shows a 0.08 point decrease above baseline, assessed up to 7 years
  Time to deterioration in quality of life, defined as the time from inclusion to the time the patient's score on the EQ-5D-3L utility score shows a 0.08 point decrease above baseline. Patients lost to follow-up without previous EQ-5D-3L deterioration will be censored at the last EQ-5D-3L assessment.
  QoL/PRO questionnaires may be filled out up until D1 every 8 weeks ±7 days during the first year, then every 12 weeks ±7 days thereafter at Progression.
PFS subgroup analysis according to Performance Status and age | From the date of first treatment administration until the date of disease progression (or death if patient died before progression), which ever occurs earlier, assessed up to 7 years
  PFS according to different subgroups :
  * PS ≥ 2 at the time of inclusion
  * Age ≥ 70 years
OS subgroup analysis according to Performance Status and age | From the date of first treatment administration until the date of death from any cause, assessed up to 7 years
  OS according to different subgroups :
  * PS ≥ 2 at the time of inclusion
  * Age ≥ 70 years
ORR subgroup analysis according to Performance Status and age | From the date of first treatment administration until the date of disease progression or death if patient died before progression) or the introduction of a new treatment, which ever occurs earlier, assessed up to 7 years
  ORR according to different subgroups :
  * PS ≥ 2 at the time of inclusion
  * Age ≥ 70 years
DCR subgroup analysis according to Performance Status and age | From the date of first treatment administration until the date of disease progression (or death if patient died before progression), which ever occurs earlier, assessed up to 7 years
  DCR according to different subgroups :
  * PS ≥ 2 at the time of inclusion
  * Age ≥ 70 years
ic-ORR subgroup analysis according to Performance Status and age | From the date of first treatment administration until the date of disease progression (or death if patient died before progression), which ever occurs earlier, assessed up to 7 years
  ic-ORR according to different subgroups :
  * PS ≥ 2 at the time of inclusion
  * Age ≥ 70 years
DOR subgroup analysis according to Performance Status and age | From the date of first documented objective response (CR or PR) until disease progression or death, which ever occurs earlier, assessed up to 7 years
  DOR according to different subgroups :
  * PS ≥ 2 at the time of inclusion
  * Age ≥ 70 years
Duration of study treatment subgroup analysis according to Performance Status and age | From the date of first treatment administration until the date of last treatment administration, up to 7 years
  Duration of treatment according to different subgroups :
  * PS ≥ 2 at the time of inclusion
  * Age ≥ 70 years
Toxicities occurring during study treatment assessed by the NCI-CTCAE v5.0, analysed in subgroups according to Performance Status and age | From the date of first treatment administration up to 30 days after the last dose of study treatment
  Proportion (%) of patients with any AE and number of events for all AEs, all SAEs and all AEs of grade ≥3 assessed by the NCI-CTCAE v5.0 criteria, according to different subgroups :
  * PS ≥ 2 at the time of inclusion
  * Age ≥ 70 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier BYLICKI, MD, PhD, PR, Study Director — HIA Sainte Anne / Groupe Français d'Onco-Pneumologie; Laurent GREILLIER, MD, PhD, PR, Study Director — AP-HM / Groupe Français d'Onco-Pneumologie
Locations (20):
- France (20):
  - CH Aix-en-Provence, Aix-en-Provence, Bouches Du Rhône
  - AP-HM, Marseille, Bouches Du Rhône
  - HIA Sainte Anne, Toulon, Var
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - Centre François Baclesse, Caen
  - CH Chambéry, Chambéry
  - Hôpitaux civils de Colmar, Colmar
  - CHI Créteil, Créteil
  - CHD Vendée, La Roche-sur-Yon
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - Hospices Civils de Lyon, Lyon
  - CH Cornouaille, Quimper
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - Hôpital Foch, Suresnes
  - CHU Toulouse, Toulouse
  - Hôpitaux Nord-Ouest, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No